CLINICAL TRIAL: NCT06336772
Title: A Comparative Trial Evaluating Restylane Shaype Versus Juvederm Volux for Chin Augmentation
Brief Title: Restylane Shaype Versus Juvederm Volux for Chin Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-2023-GAL-SHYP
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Chin Retrusion
Keywords: Chin Augmentation; Hyaluronic Acid Filler; Aesthetic Injection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Shaype (Experimental): Restylane Shaype is approved and commercially available for use in Canada and is manufactured by Q-Med AB, part of the Galderma Group.
  The participant will be treated at the Baseline visit and will be eligible for retreatment 2 weeks later if a touch up is deemed necessary by the Treating Investigator. Volumes used for each participant will be determined by the aesthetic judgement of the Treating Investigator.
  Interventions: Device: Restylane Shaype
- Juvederm Volux (Active Comparator): Juvéderm Volux is approved and commercially available for use in Canada and is manufactured by Allergan Aesthetics, an Abbvie company.
  The participant will be treated at the Baseline visit and will be eligible for retreatment 2 weeks later if a touch up is deemed necessary by the Treating Investigator. Volumes used for each participant will be determined by the aesthetic judgement of the Treating Investigator.
  Interventions: Device: Juvéderm Volux

INTERVENTIONS:
Device: Restylane Shaype — Half (50%) of study participants will receive Restylane Shaype for the treatment of mild to severe chin retrusion
  Arms: Restylane Shaype
Device: Juvéderm Volux — Half (50%) of study participants will receive Juvéderm Volux for the treatment of mild to severe chin retrusion
  Arms: Juvederm Volux

SUMMARY:
This study aims to compare two injectable products (Restylane Shaype and Juvéderm Volux) for aesthetic augmentation of the chin

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, male and female subjects 18 years of age and older.
2. Patients with established chin retrusion at Baseline (a score of mild, moderate, and severe severity on the Galderma Chin Retrusion Scale).
3. Accepted the obligation not to receive any other facial procedures throughout the study duration.
4. Understood and accepted the obligation and would be logistically able to appear for all scheduled follow-up visits.
5. No previous lower face fillers for 12 months prior to this study.
6. Capable of providing informed consent.

Exclusion Criteria:

1. Patients without chin retrusion at Baseline, per the Galderma Chin Retrusion Scale.
2. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)].
3. Hypersensitivity to Restylane or Juvéderm products, hyaluronic acid filler or amide local anesthetics.
4. Patients presenting with porphyria or any other liver diseases.
5. Inability to comply with follow-up and abstain from facial injections during the study period.
6. Heavy smokers, classified as smoking more than 12 cigarettes per day.
7. History of severe or multiple allergies manifested by anaphylaxis since drug allergies might preclude optimal management of complications.
8. Previous tissue revitalization therapy in the treatment area (i.e., the lower face) within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion.
9. Previous facial surgery, including liposuction.
10. Lifetime history of permanent implants in the treatment region (i.e., the lower face)
11. Lifetime history of semi-permanent dermal fillers in the treatment region (i.e., the lower face).
12. History or presence of any disease or lesion near or at the treatment area, including inflammation, active or chronic infection, including in the mouth, dentals, head, and neck region.
13. Active facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes zoster or any other facial condition that may increase the risk of cutaneous penetration of infective agents.
14. Scars, deformities, piercings, or tattoos in the treatment areas.
15. Facial cancer or precancer (e.g., actinic keratosis).
16. History of radiation therapy in the treatment area.
17. History of bleeding disorders, or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g., Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment.
18. Patients with immune disorders such as systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, and Hashimoto's thyroiditis, or subjects using immunosuppressants.
19. Patients with a tendency to form hypertrophic or keloid scars, or any other healing disorders.
20. Patients with a tendency to form post-inflammatory hyperpigmentation.
21. Patients with known hypersensitivity to lidocaine or agents structurally related to amide type local anesthetics (e.g., certain anti-arrhythmics).
22. Patients administered dental block or topical administration of lidocaine within 2 weeks of treatment.
23. Patients with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction.
24. Current remote infections (e.g., urinary tract, sinuses, intestinal tract, oral cavity)
25. Planned dental procedures during the 2-week period before and after filler treatments, including teeth cleaning, tooth extraction and gum grafts.
26. Planned COVID-19 vaccinations during the 2-week period before and after filler treatments.
27. Lifetime history of cystic acne, due to increased risk of cyst development following filler treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Statistically significant group differences in the average three-dimensional volumetric increase since baseline | Baseline to Week 2, Week 4, Week 12, Week 24
  As assessed by the Canfield Vectra XT system.

SECONDARY OUTCOMES:
Treatment group differences assessed by blinded evaluations on a validated chin retrusion scale (Galderma Chin Retrusion Scale) | Baseline to Week 2, Week 4, Week 12, Week 24
  The Galderma Chin Retrusion Scale is a 4 point Likert Scale used to assess chin retrusion ranging from "no retrusion" (grade 0) to "severe retrusion" (grade 3)
Treatment group differences assessed by blinded evaluations of aesthetic improvement (Global Aesthetic Improvement Scale) | Baseline to Week 2, Week 4, Week 12, Week 24
  The Global Aesthetic Improvement Scale is a 5 point Likert Scale in which the blinded investigator can assess change in chin retrusion following aesthetic treatment. The grading scale ranges from "worse" (grade -1) to "very much improved" (grade 3)
Assessment of product integration by means of ultrasound (the radius or surface area of in vivo product placed within tissues, integration [or lack thereof] of the product into the surrounding tissues) | Baseline to Week 2, Week 4, Week 12, Week 24
  This will be done by means of measurement of the radius or surface area of in vivo product placed within tissues, integration [or lack thereof] of the product into the surrounding tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No